CLINICAL TRIAL: NCT01268202
Title: Curative Efficacy of Pravastatine in Patients Presented Delayed Cutaneous and Subcutaneous Radio-induced Fibrosis
Acronym: PRAVACUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSET 1383 - PRAVACUR
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Fibrosis
Keywords: cutaneous radioinduced fibrosis
MeSH Terms: conditions — Fibrosis | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pravastatin (Experimental): Pravastatin : 40mg/day during 12 months
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Pravastatin 40mg/day during 12 months

SUMMARY:
Molecular mechanisms involved in radio-induced fibrosis are assessed in UPRES EA 27-10 since 10 years. Besides the canonical TGFbeta/ Smad pathway involved in radio-induced fibrosis (RIF), the Rho/ROCK/CTGF cascade has been shown to be also implicated in molecular mechanisms of RIF. Curative administration of Pravastatin or ROCK specific inhibitors inhibits the chronically activated Rho/ROCK/CTGF pathway in vitro in human cells lines and ex vivo in human samples. In addition, the curative administration of Pravastatin improves established RIF in vivo. The investigators data suggest that the pravastatin-based strategy is an efficient and safe antifibrotic therapy, easily transferable into the clinic to improve the quality of life of long-term cancer survivors without interfering with prior anticancer treatment.

This clinical trial evaluates the curative efficacy of Pravastatine in patients who presented a cutaneous and/ or subcutaneous fibrosis (grade >= 2 according to NCI-CTCAE v4 toxicities scale) and who were treated by radiotherapy for a head and neck cancer. Patients will be treated by Pravastatin during 12 months. An intermediate evaluation of efficacy by ultrasound will be assessed at 6 months and at last, at the end of the treatment. Patients assessment will be performed at 6 and 12 months after the end of the treatment to look at a potential rebound effect.

Objective(s) of the clinical study

Main objective: To assess Pravastatin efficacy in established cutaneous and subcutaneous radio-induced fibrosis revealed from 6 to 24 months after head and neck radiotherapy.

Second objective: To evaluate radio-induced fibrosis regression during the year following treatment stop.

ELIGIBILITY:
Inclusion Criteria:

1. Grade >= 2 cutaneous and/or subcutaneous fibrosis (NCI-CTCAE v4 toxicities scale) revealed from 6 to 24 months after head and neck radiotherapy.
2. Head and neck cancers treated by radiation therapy +/- chemotherapy, +/- surgery, with no evidence of progressive disease.
3. Age >= 18
4. Karnofsky PS ≥ 70
5. normal renal function (plasmatic creatinine <= 130 micromol/l), normal cholesterol, normal hepatic function (total bilirubin <= 1.5 UNL, SGOT and SGPT <= 2 UNL)
6. Written informed consent of the patient.

Exclusion Criteria:

1. any chronic treatment by corticoids
2. severe cardiac pathology
3. patients already treated by statins or treated by fibrates, cyclosporine
4. history of muscular toxicities when treated by fibrates or by statins
5. Personal or familial history of hereditary muscular pathology
6. Plasmatic CPK >3 UNL
7. patient already included in another therapeutic trial with an experimental drug,
8. pregnant patient or susceptible to pregnancy or breast feeding (patients in age to give birth must be placed under efficient contraception),
9. a social or psychological condition that does not allow a positive patient's participation in the treatment and necessary medical follow-up to be envisaged,
10. the patient is under legal restrained or tutelage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-12-17 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
regression of radio-induced fibrosis (RIF) evaluated by high frequency ultrasound | 12 months
  a decrease of the maximal thickness more than 30% compared to RIF before treatment.

SECONDARY OUTCOMES:
Fibrosis grade according to NCI-CTCAE v4 toxicities scale. | 12 months
Quality of life | 12 months
  VQ-Dermato scale

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Rivera, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (3):
- France (3):
  - Centre Val d'Aurelle, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Bourgier C, Auperin A, Rivera S, Boisselier P, Petit B, Lang P, Lassau N, Taourel P, Tetreau R, Azria D, Bourhis J, Deutsch E, Vozenin MC. Pravastatin Reverses Established Radiation-Induced Cutaneous and Subcutaneous Fibrosis in Patients With Head and Neck Cancer: Results of the Biology-Driven Phase 2 Clinical Trial Pravacur. Int J Radiat Oncol Biol Phys. 2019 Jun 1;104(2):365-373. doi: 10.1016/j.ijrobp.2019.02.024. Epub 2019 Feb 15. PMID 30776452
- See also: Institut Gustave Roussy — http://igr.fr